CLINICAL TRIAL: NCT03809260
Title: A Clinical Trial for Analysis of Intestinal Microbiome Affecting Pharmacokinetics, Pharmacodynamics, and Safety of Metformin in Healthy Volunteers
Brief Title: A Clinical Trial for Analysis of Intestinal Microbiome Affecting PK, PD, and Safety of Metformin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, MD, PhD, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MMP
Record Dates: First submitted 2019-01-08; First posted 2019-01-18 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Human Microbiome
MeSH Terms: interventions — Metformin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 (Experimental): Metformin/Vancomycin
  Interventions: Drug: Metformin (part 1); Drug: Vancomycin
- Part 2 (Experimental): Metformin
  Interventions: Drug: Metformin (part 2)

INTERVENTIONS:
Drug: Metformin (part 1) — 1~4d: Metformin 1000 mg bid (Except for 500 mg after 1d lunch), 16d~19d: Metformin 1000 mg bid (Except for 500 mg after 16d lunch).
  Other Names: Diabex Tab., 500 mg
  Arms: Part 1
Drug: Vancomycin — 11d: Vancomycin 250 mg bid, 12~17d: Vancomycin 500 mg bid
  Other Names: Vancozin cap., 250 mg
  Arms: Part 1
Drug: Metformin (part 2) — 1~4d: Metformin 1000 mg bid (Except for 500 mg after 1d lunch)
  Other Names: Diabex Tab., 500 mg
  Arms: Part 2

SUMMARY:
This clinical trial is intended to evaluate the effects of the changes in intestinal microbiome by antibiotics (PO vancomycin) on the pharmacokinetic /pharmacodynamic and safety profiles of metformin in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 45, healthy male subjects(at screening)
* Body weight between 50.0 kg - 100.0 kg, BMI between 18.0 - 28.0 kg/m2
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Subject who has a past or present history of any diseases following below.(liver, kidney, neurology, immunology, pulmonary, endocrine, hematology, oncology, cardiology, mental disorder)
* Subject who had GI tract disease(Crohn's disease, ulcer, acute or chronic pancreatitis) or surgery (appendectomy, hernioplasty are excluded)
* Serum AST(SGOT), ALT(SGPT)>1.5 times upper limit of normal range
* MDRD eGFR <80mL/min/1.73m2
* Subject who had drug (Aspirin, antibiotics) hypersensitivity reaction
* Subject who already participated in other trials in 3 months
* Subject who had whole blood donation in 2 months, or component blood donation in 1 month or transfusion in 1 month currently.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Compare the gut microbiome species change | Day 1/4/16/19
  Compare how the gut microbiome species change after metformin (or vancomycin) multiple dosing

SECONDARY OUTCOMES:
Compare the maximum plasma concentration (Cmax) of metformin | Day 4/19 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours post-dose)
  Compare the maximum plasma concentration (Cmax) of metformin before and after vancomycin PO treatment
Compare the area under the plasma concentration versus time curve (AUC) of metformin | Day 4/19 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours post-dose)
  Compare the area under the plasma concentration versus time curve (AUC) of metformin before and after vancomycin PO treatment
Compare the maximum blood glucose concentration (Gmax) | Day 1/4/16/19 (pre-dose (75 g glucose), 0.25, 0.5, 0.75, 1, 1.5. 2 hours)
  Oral glucose tolerance test (OGTT); Compare the maximum blood glucose concentration (Gmax) before and after metformin (or vancomycin) PO treatment
Compare the area under the blood glucose concentration versus time curve (AUC) | Day 1/4/16/19 (pre-dose (75 g glucose), 0.25, 0.5, 0.75, 1, 1.5. 2 hours)
  Oral glucose tolerance test (OGTT); Compare the area under the blood glucose concentration versus time curve (AUC) before and after metformin (or vancomycin) PO treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- SNUBH Clinical trial centor, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim E, Kim AH, Lee Y, Ji SC, Cho JY, Yu KS, Chung JY. Effects of vancomycin-induced gut microbiome alteration on the pharmacodynamics of metformin in healthy male subjects. Clin Transl Sci. 2021 Sep;14(5):1955-1966. doi: 10.1111/cts.13051. Epub 2021 May 31. PMID 33982376